CLINICAL TRIAL: NCT02068885
Title: Dietary Composition and Energy Expenditure During Weight-Loss Maintenance
Brief Title: Framingham State Food Study
Acronym: (FS)2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Framingham State University (Other); Baylor College of Medicine (Other); Nutrition Science Initiative (Other); New Balance Foundation (Other); Many Voices Foundation (Other); Blue Cross Blue Shield (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Director, Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00009571
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Diabetes; Cardiovascular Disease
Keywords: Low carbohydrate diet; Low fat diet; Glycemic index; Weight loss maintenance
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low carbohydrate diet (Experimental): Feeding study. Composition (by proportion of calories): 20% carbohydrate, 60% fat, 20% protein
  Interventions: Behavioral: Feeding study
- Moderate carbohydrate diet (Experimental): Feeding study. Composition (by proportion of calories): 40% carbohydrate, 40% fat, 20% protein
  Interventions: Behavioral: Feeding study
- High carbohydrate diet (Active Comparator): Feeding study. Composition (by proportion of calories): 60% carbohydrate, 20% fat, 20% protein
  Interventions: Behavioral: Feeding study

INTERVENTIONS:
Behavioral: Feeding study — Food provision throughout the study to all 3 dietary arms, with the following phases: 1) Weight loss; 2) Weight maintenance; 3) Ad libitum

SUMMARY:
This study will evaluate the effects of dietary composition on energy expenditure and chronic disease risk factors, while also exploring physiological mechanisms underlying these effects.

DETAILED DESCRIPTION:
Many overweight and obese people can lose weight for a few months, but most have difficulty maintaining weight loss over the long term. One explanation for the poor long-term outcome of weight-loss diets relates to behavior, in that motivation to adhere to restrictive regimens typically diminishes with time. An alternative explanation is that weight loss elicits biological adaptations - specifically a decline in energy expenditure and an increase in hunger - that promote weight regain. The purpose of this study is to evaluate the effects of dietary composition on energy expenditure and risk for chronic diseases, while also exploring physiological mechanisms underlying these effects. The study will be performed in collaboration with Framingham State University, providing a novel and feasible method for feeding subjects in dining halls and monitoring compliance.

Following 12±2% weight loss on a standard run-in diet, 150 adults (aged 18 to 65 years) will be randomly assigned to one of three weight-loss maintenance diets controlled for protein content (20% of energy) and varying widely in dietary carbohydrate-to-fat ratio: Low-carbohydrate (20% of energy from carbohydrate, 60% fat), Moderate- carbohydrate (40% carbohydrate, 40% fat), High-carbohydrate (60% carbohydrate, 20% fat). During the weight-loss maintenance phase, energy intake will be adjusted to prevent changes in body weight. The primary outcome will be change in total energy expenditure (indirect calorimetry using stable isotopes) through 20 weeks. Secondary outcomes during weight maintenance will include resting energy expenditure (indirect calorimetry using respiratory gas exchange), physical activity (accelerometry), measures of insulin resistance and skeletal muscle work efficiency, components of the metabolic syndrome, and hormonal and metabolic measures that might inform an understanding of physiological mechanisms. We also will assess weight change during a 2-week ad libitum feeding phase, as an objective measure of dietary effects on hunger. The analytic framework for addressing study hypothesis will be repeated-measures analysis of variance, with adjustment for covariates (sex, race, ethnicity, age, anthropometrics, insulin sensitivity and secretion, obesity-related genes). We also will test each covariate for effect modification (covariate × diet interaction).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* BMI ≥ 25 kg/m2
* Weight ≤ 425 lbs
* Medical clearance from a primary care provider
* Plans to matriculate at Framingham State University (campus-based participants: students), work on campus (campus-based participants: faculty and staff), or live in the greater Framingham area (community-based participants) throughout the academic year of enrollment in the study
* Academic and social clearance from the FSU Office of Enrollment and Student Development (student participants) or willingness to comply with Criminal Offender Record Information (CORI) check and Sex Offender Registry Information (SORI) check (community-based subjects)
* Willingness to eat and drink only the foods and beverages on the study menus during participation, with no food allergies or aversions
* Willingness to eat in the dining hall
* Willingness to abstain from consuming alcohol during participation

Exclusion Criteria:

* Change in body weight exceeding ±10% during prior year
* Recent adherence to a special diet
* Recent adherence to a vigorous physical activity regimen (e.g., participation in a varsity sport)
* Chronic use of any medication or dietary supplement that could affect study outcomes
* Current smoking (1 cigarette in the last week)
* Heavy baseline alcohol consumption (> 10 drinks/week) or history of binge drinking (≥ 5 drinks in 1 day, anytime in past 6 months)
* Physician diagnosis of a major medical/psychiatric illness or eating disorder
* Abnormal HgA1c, TSH, BUN, creatinine; hematocrit < 30; ALT > 200% of normal upper limit
* Plans for a vacation during the study that would preclude adherence to prescribed diet
* Additional exclusions for female participants: Irregular menstrual cycles; any change in birth control medication during the 3 months prior to enrollment; pregnancy or lactation during the 12 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2014-08-17 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Klein, MS, RD, Study Director — Boston Children's Hospital; Cara B Ebbeling, PhD, Principal Investigator — Boston Children's Hospital; David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Framingham State University, Framingham, Massachusetts, United States

REFERENCES:
- [Background] Wong JM, Bielak L, Eddy RG, Stone L, Lakin PR, Sandman M, Devlin C, Seger-Shippee L, Wiroll D, Luoto PK, Klein GL, Ludwig DS, Ebbeling CB. An Academia-Industry Partnership for Planning and Executing a Community-Based Feeding Study. Curr Dev Nutr. 2018 Jul 5;2(9):nzy060. doi: 10.1093/cdn/nzy060. eCollection 2018 Sep. PMID 30283914
- [Background] Ebbeling CB, Klein GL, Luoto PK, Wong JMW, Bielak L, Eddy RG, Steltz SK, Devlin C, Sandman M, Hron B, Shimy K, Heymsfield SB, Wolfe RR, Wong WW, Feldman HA, Ludwig DS. A randomized study of dietary composition during weight-loss maintenance: Rationale, study design, intervention, and assessment. Contemp Clin Trials. 2018 Feb;65:76-86. doi: 10.1016/j.cct.2017.12.004. Epub 2017 Dec 9. PMID 29233719
- [Background] Ludwig DS, Greco KF, Ma C, Ebbeling CB. Testing the carbohydrate-insulin model of obesity in a 5-month feeding study: the perils of post-hoc participant exclusions. Eur J Clin Nutr. 2020 Jul;74(7):1109-1112. doi: 10.1038/s41430-020-0658-8. Epub 2020 May 20. PMID 32435054
- [Result] Ebbeling CB, Feldman HA, Klein GL, Wong JMW, Bielak L, Steltz SK, Luoto PK, Wolfe RR, Wong WW, Ludwig DS. Effects of a low carbohydrate diet on energy expenditure during weight loss maintenance: randomized trial. BMJ. 2018 Nov 14;363:k4583. doi: 10.1136/bmj.k4583. PMID 30429127
- [Result] Ebbeling CB, Bielak L, Lakin PR, Klein GL, Wong JMW, Luoto PK, Wong WW, Ludwig DS. Energy Requirement Is Higher During Weight-Loss Maintenance in Adults Consuming a Low- Compared with High-Carbohydrate Diet. J Nutr. 2020 Aug 1;150(8):2009-2015. doi: 10.1093/jn/nxaa150. PMID 32470981
- [Derived] Angelidi AM, Bartell E, Huang Y, Zeleznik OA, Estanyol-Torres N, Mi MY, Bhupathiraju SN, Kelly RS, Wittenbecher C, Lasky-Su J, Clish CB, Ludwig DS, Ebbeling CB, Hirschhorn JN. Weight-independent effects of dietary carbohydrate-to-fat ratio on metabolomic profiles: secondary outcomes of a 5-month randomized controlled feeding trial. Nat Commun. 2026 Jan 17. doi: 10.1038/s41467-026-68353-z. Online ahead of print. PMID 41547934
- [Derived] Wong JMW, Yu S, Ma C, Mehta T, Dickinson SL, Allison DB, Heymsfield SB, Ebbeling CB, Ludwig DS. Stimulated Insulin Secretion Predicts Changes in Body Composition Following Weight Loss in Adults with High BMI. J Nutr. 2022 Mar 3;152(3):655-662. doi: 10.1093/jn/nxab315. PMID 34587231
- [Derived] Ebbeling CB, Knapp A, Johnson A, Wong JMW, Greco KF, Ma C, Mora S, Ludwig DS. Effects of a low-carbohydrate diet on insulin-resistant dyslipoproteinemia-a randomized controlled feeding trial. Am J Clin Nutr. 2022 Jan 11;115(1):154-162. doi: 10.1093/ajcn/nqab287. PMID 34582545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants by posting flyers, newspaper advertisements, and Internet announcements.
Pre-assignment Details: We enrolled 234 participants for the run-in phase. Of these, 164 participants achieved at least 10% weight loss and were randomly assigned to one of three diets for the test phase (low-carbohydrate diet, n=57; moderate-carbohydrate diet, n=53; or high-carbohydrate diet, n=54).
Period: Overall Study
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Started (Sample size randomized) | 57 | 53 | 54
Provided data at midpoint test phase | 56 | 50 | 48
Provided data at end of test phase (Sample size completers) | 54 | 48 | 46
Included in intention-to-treat analysis (Two randomized participants excluded: unreliable doubly labeled water (DLW) data, hypothyroidism) | 56 | 52 | 54
Completed | 54 | 48 | 46
Not Completed | 3 | 5 | 8
Not completed — Withdrew | 3 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet | Total
Number analyzed (Participants) | 57 | 53 | 54 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 53 | 54 | 164
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — pre-weight loss, beginning of run-in phase
  years | 37.1 (13.3) | 37.3 (14.9) | 39.8 (15.1) | 37.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 42 | 115
  Male | 20 | 17 | 12 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 8 | 25
  Not Hispanic or Latino | 47 | 46 | 46 | 139
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 53 | 54 | 164
Total Energy Expenditure [Mean (Standard Deviation); unit: kcal/d] — pre-weight loss, beginning of run-in phase
  kcal/d | 3110 (680) | 3030 (788) | 2915 (686) | 3021 (719)

OUTCOME MEASURES:

1. Primary Outcome: Total Energy Expenditure, Assessed by Indirect Calorimetry Using Stable Isotopes
Description: Total energy expenditure (TEE), assessed by indirect calorimetry using stable isotopes
  Total calories burned: Participants each drank about a cup of water containing special tracers which are measurable when they pass out of the body through urine. They provided a urine sample before they drank the water and then about every other day for the next two (2) weeks.
  Change: average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Start of Trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: kcal/d
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 52 | 54
kcal/d
  Start of Trial | 2713 [2696 to 2730] | 2504 [2486 to 2522] | 2640 [2623 to 2657]
  Change | 190 [109 to 270] | 71 [-12 to 155] | -19 [-104 to 66]

2. Secondary Outcome: Resting Energy Expenditure, Assessed by Indirect Calorimetry Using Respiratory Gas Exchange
Description: Resting energy expenditure, assessed by indirect calorimetry using respiratory gas exchange Calories burned while resting: Participants lied down with head and neck under a clear plastic "bubble," breathing room air. Gases in expired air were collected.
  Change: average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: kcal/d
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
kcal/d
  Start of Trial | 1615 [1609 to 1621] | 1576 [1569 to 1583] | 1603 [1597 to 1609]
  Change | 54 [32 to 76] | 46 [23 to 69] | 34 [10 to 57]

3. Secondary Outcome: Physical Activity, Assessed by Accelerometry
Description: Actigraph Accelerometer Change: average (midpoint of test phase, end of test phase) - start of trial An Actigraph Accelerometer measures movement, similar to a pedometer. Data are reported as counts (divided by 1,000) per day. Each participant wore the the accelerometer on the right hip for 7 days at each time point.
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: counts/d
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 55 | 52 | 54
counts/d
  Start of Trial | 495.8 [489.5 to 502.1] | 463.8 [457.0 to 470.6] | 476.6 [470.4 to 482.8]
  Change | -6.9 [-31.0 to 17.1] | -42.4 [-67.7 to -17.1] | -26.3 [-52.0 to -0.6]

4. Secondary Outcome: Skeletal Muscle Work Efficiency
Description: Efficiency is expressed as percentage ratio of power generated during cycle ergometry (with conversion of Watts to kcal/min using a factor of 0.01433) to energy expenditure above resting.
  Change: end of test phase - start of trial.
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Measure: Mean (95% Confidence Interval); unit: % power generated to energy expended
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 55 | 51 | 53
% power generated to energy expended
  Start of Trial | 12.2 [12.1 to 12.3] | 11.7 [11.6 to 11.8] | 12.2 [12.1 to 12.3]
  Change | 0.3 [-0.3 to 0.9] | -0.0 [-0.6 to 0.6] | -0.1 [-0.8 to 0.5]

5. Secondary Outcome: Leptin (Start of Trial)
Description: Leptin levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units (exp(mean log)±exp(mean log)×(exp(SE log)-1)).
  Changes (see Outcome 6) are expressed in percentage units (100%×(exp(change in log)-1)): average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
ng/mL | 9.6 [9.2 to 10.0] | 9.8 [9.4 to 10.2] | 10.9 [10.5 to 11.3]

6. Secondary Outcome: Leptin (% Change)
Description: Leptin levels were log transformed for analysis. Change (expressed in percentage units, 100%×(exp(change in log)-1)): average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Change through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
% change | 17.9 [7.7 to 29.1] | 34.8 [22.6 to 48.2] | 34.2 [21.8 to 47.7]

7. Secondary Outcome: Ghrelin (Start of Trial)
Description: Ghrelin levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units (exp(mean log)±exp(mean log)×(exp(SE log)-1)).
  Changes (see Outcome 8) are expressed in percentage units (100%×(exp(change in log)-1)): average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
pg/mL | 598.2 [586.3 to 610.1] | 640.1 [626.4 to 653.8] | 693.2 [679.5 to 706.9]

8. Secondary Outcome: Ghrelin (% Change)
Description: Ghrelin levels were log transformed for analysis. Change (expressed in percentage units, 100%×(exp(change in log)-1)): average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Change through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
% change | -11.8 [-14.8 to -8.6] | -8.7 [-12.0 to -5.3] | -4.9 [-8.4 to -1.2]

9. Secondary Outcome: 1,5-Anhydroglucitol
Description: Biomeasure of carbohydrate intake Change, 10 weeks: midpoint of test phase - start of trial Change, 20 weeks: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
ug/mL
  Start of Trial | 16.7 [16.2 to 17.2] | 17.2 [16.7 to 17.7] | 17.1 [16.7 to 17.6]
  Change, 10 weeks | -2.5 [-3.0 to -2.0] | -1.2 [-1.7 to -0.7] | 0.1 [-0.4 to 0.6]
  Change, 20 weeks | -3.5 [-4.2 to -2.8] | -1.8 [-2.6 to -1.1] | 0.6 [-0.2 to 1.3]

10. Secondary Outcome: Glycemic Control, Assessed by HgA1c
Description: Change, 10 weeks: midpoint of test phase - start of trial. Change, 20 weeks: end of test phase - start of trial.
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Measure: Mean (95% Confidence Interval); unit: % hemoglobin with glucose bound
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
% hemoglobin with glucose bound
  Start of Trial | 5.56 [5.52 to 5.60] | 5.58 [5.54 to 5.62] | 5.61 [5.57 to 5.65]
  Change, 10 weeks | 0.01 [-0.02 to 0.04] | 0.03 [0.00 to 0.06] | -0.01 [-0.05 to 0.02]
  Change, 20 weeks | -0.01 [-0.04 to 0.03] | 0.00 [-0.03 to 0.04] | -0.05 [-0.08 to -0.01]

11. Secondary Outcome: Triglycerides
Description: Triglyceride levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units Change, 10 weeks: midpoint of test phase - start of trial Change, 20 weeks: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Measure: Mean (95% Confidence Interval); unit: md/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
md/dL
  Start of Trial | 77.3 [71.1 to 84.0] | 76.5 [70.2 to 83.3] | 80.5 [74.2 to 87.4]
  Change, 10 weeks | -12.1 [-18.5 to -5.1] | 8.4 [0.0 to 17.5] | 10.9 [2.3 to 20.2]
  Change, 20 weeks | -12.8 [-19.8 to -5.2] | -0.1 [-8.5 to 9.1] | 7.5 [-1.7 to 17.6]

12. Secondary Outcome: Body Composition (DXA)
Description: Body fat, presented as a % of total mass
  Participants each had a special scan (x-ray) to measure their amount of body fat. The special x-ray is called "dual-energy x-ray absorptiometry" (DXA). They were asked to lie still on a table for x-ray pictures.
  Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: % of total body mass
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 52 | 54
% of total body mass
  Start of Trial | 36.2 [34.6 to 37.9] | 37.3 [35.1 to 39.5] | 37.8 [36.2 to 39.4]
  Change | -0.3 [-0.7 to 0.2] | -0.3 [-0.7 to 0.1] | -0.5 [-1.0 to -0.1]

13. Secondary Outcome: Glucose
Description: Glucose level, fasting blood draw Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Intention-to-treat analysis
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 52 | 54
mg/dL
  Start of Trial | 95.1 [92.9 to 97.2] | 94.3 [91.9 to 96.8] | 95.1 [92.9 to 97.3]
  Change | 1.0 [-0.9 to 2.8] | -0.3 [-2.2 to 1.7] | -1.0 [-3.0 to 0.9]

14. Secondary Outcome: Change in Lipoprotein Particle Subfraction Distribution
Description: Lipoprotein insulin resistance (LPIR) score was calculated from triglyceride-rich, high-density, and low-density lipoprotein particle (TRL-P, HDL-P, LDL-P) sizes and subfraction concentrations (large/very large TRL-P, large HDL-P, small LDL-P). LPIR score is quantified on a scale of 0-100. Higher scores indicate worse outcome.
  Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Retention rate was 90%, with 148 of 164 participants completing the study and 147 included in the analysis (after a priori exclusion of one participant who developed hypothyroidism).
Measure: Mean (95% Confidence Interval); unit: score on a scale (0-100)
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
score on a scale (0-100)
  Start of trial | 34.6 [28.7 to 40.5] | 31.5 [26.1 to 36.9] | 31.4 [26.9 to 35.9]
  Change | -5.3 [-9.2 to -1.5] | -0.02 [-4.1 to 4.1] | 3.6 [-0.6 to 7.7]

15. Secondary Outcome: Total Cholesterol
Description: Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
mg/dL
  Start of trial | 147.5 [140.2 to 154.9] | 145.5 [136.1 to 154.8] | 142.9 [135.1 to 150.8]
  Change | 16.1 [11.5 to 20.7] | 18.5 [13.6 to 23.3] | 16.2 [11.2 to 21.1]

16. Secondary Outcome: HDL-Cholesterol
Description: High-density lipoprotein cholesterol Change, 10 weeks: midpoint of test phase - start of trial. Change, 20 weeks: end of test phase - start of trial.
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Measure: Mean (95% Confidence Interval); unit: md/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 51 | 54
md/dL
  Start of Trial | 47.8 [45.7 to 49.8] | 49.1 [47.0 to 51.2] | 47.6 [45.5 to 49.6]
  Change, 10 weeks | 11.1 [9.4 to 12.8] | 6.9 [5.1 to 8.7] | 4.7 [2.9 to 6.5]
  Change, 20 weeks | 13.0 [11.0 to 15.0] | 9.7 [7.6 to 11.8] | 6.8 [4.7 to 8.9]

17. Secondary Outcome: Non-HDL-Cholesterol
Description: Calculated by subtracting HDL-cholesterol from total cholesterol. Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (97.5% Confidence Interval); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
mg/dL
  Start of trial | 101.5 [94.1 to 108.9] | 99.0 [90.6 to 107.5] | 98.2 [91.2 to 105.3]
  Change | 6.3 [1.8 to 10.9] | 11.0 [6.3 to 15.8] | 9.5 [4.6 to 14.4]

18. Secondary Outcome: LDL-Cholesterol
Description: Low-density-lipoprotein cholesterol Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
mg/dL
  Start of trial | 80.6 [75.1 to 86.1] | 77.6 [70.3 to 84.9] | 79.5 [73.2 to 85.8]
  Change | 10.0 [6.3 to 13.7] | 11.7 [7.8 to 15.7] | 8.2 [4.2 to 12.2]

19. Secondary Outcome: Adiponectin (Start of Trial)
Description: Total and high molecular weight adiponectin Adiponectin levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units (exp(mean log)±exp(mean log)×(exp(SE log)-1)).
  Changes (see Outcome 20) are expressed in percentage units (100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
ng/mL
  Total | 4.0 [3.0 to 5.9] | 5.1 [3.3 to 7.2] | 4.9 [3.5 to 5.9]
  High Molecular Weight | 2.3 [1.4 to 3.5] | 2.8 [1.6 to 4.2] | 2.7 [1.9 to 3.6]

20. Secondary Outcome: Adiponectin (% Change)
Description: Adiponeptin levels were log transformed for analysis. Change (expressed in percentage units, 100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Change through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
% change
  Total | 33.6 [24.9 to 42.9] | 17.4 [9.4 to 26.0] | 23.0 [14.5 to 32.3]
  High Molecular Weight | 42.9 [33.3 to 53.1] | 27.6 [18.6 to 37.2] | 27.8 [18.7 to 37.7]

21. Secondary Outcome: C-reactive Protein (Start of Trial)
Description: C-reactive protein, marker of inflammation C-reactive protein levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units (exp(mean log)±exp(mean log)×(exp(SE log)-1)).
  Changes (see Outcome 22) are expressed in percentage units (100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
mg/L | 1.1 [0.6 to 2.5] | 1.5 [0.7 to 4.6] | 1.5 [0.6 to 3.1]

22. Secondary Outcome: C-reactive Protein (% Change)
Description: C-reactive protein, marker of inflammation C-reactive protein levels were log transformed for analysis. Change (expressed in percentage units, 100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Change through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
% change | -9.9 [-24.2 to 7.1] | -20.6 [-33.8 to -4.8] | -1.7 [-18.6 to 18.6]

23. Secondary Outcome: IL-6 (Start of Trial)
Description: Interleukin-6, marker of inflammation Interleukin-6 levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units (exp(mean log)±exp(mean log)×(exp(SE log)-1)).
  Changes (see Outcome 24) are expressed in percentage units (100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
pg/mL | 1.4 [1.0 to 2.4] | 1.8 [1.1 to 3.3] | 1.7 [1.0 to 2.6]

24. Secondary Outcome: IL-6 (% Change)
Description: Interleukin-6, marker of inflammation Interleukin-6 levels were log transformed for analysis. Change (expressed in percentage units, 100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Change through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
% change | -23.6 [-35.4 to -9.6] | -20.1 [-33.0 to -4.7] | -18.3 [-31.8 to -2.2]

25. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
mmHg
  Systolic, Start of trial | 117.2 [114.7 to 119.7] | 119.2 [115.9 to 122.5] | 114.3 [111.8 to 116.9]
  Systolic, Change | -1.5 [-4.4 to 1.5] | 0.0 [-3.1 to 3.1] | 1.8 [-1.3 to 5.0]
  Diastolic, Start of trial | 70.7 [68.3 to 73.1] | 73.7 [71.3 to 76.0] | 70.5 [68.3 to 72.7]
  Diastolic, Change | 2.2 [-0.4 to 4.8] | 1.4 [-1.3 to 4.1] | 2.2 [-0.6 to 5.0]

26. Secondary Outcome: Plasminogen Activator Inhibitor-1 (Start of Trial)
Description: Plasminogen activator inhibitor-1 levels were log transformed for analysis. For reporting, the adjusted means and 95% Confidence Intervals were retransformed to the original units (exp(mean log)±exp(mean log)×(exp(SE log)-1)).
  Changes (see Outcome 27) are expressed in percentage units (100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
ng/mL | 1.1 [0.7 to 2.5] | 1.5 [0.7 to 3.1] | 1.2 [0.6 to 2.1]

27. Secondary Outcome: Plasminogen Activator Inhibitor-1 (% Change)
Description: Plasminogen activator inhibitor-1 levels were log transformed for analysis. Change (expressed in percentage units, 100%×(exp(change in log)-1)): end of test phase - start of trial
Time Frame: Change through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
% change | 7.2 [-14.7 to 34.8] | 26.9 [-0.2 to 61.4] | 14.9 [-10.1 to 46.9]

28. Secondary Outcome: Fibrinogen
Description: Change: end of test phase - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: as for outcome 14
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 53 | 48 | 46
mg/dL
  Start of trial | 421.1 [398.2 to 443.9] | 461.0 [430.7 to 491.4] | 428.1 [400.9 to 455.2]
  Change | -17.0 [-36.8 to 2.7] | -22.4 [-43.2 to -1.7] | -21.7 [-42.9 to -0.5]

29. Secondary Outcome: Insulin Secretion Determined as Blood Insulin Concentration 30 Minutes After Oral Glucose (Start of Trial)
Description: Insulin level 30 minutes after consuming 75 grams of glucose
Time Frame: Start of trial (time of randomization, post-weight loss)
Population: Descriptive data, reflecting participant flow Pre-weight loss (N=162, minus 1 participant in the Moderate carbohydrate diet group for whom insulin-30 result is missing) Start of trial (N=162) End of test phase (N=148, minus 1 participant in the High carbohydrate diet group for whom insulin-30 result is missing)
Measure: Median (Inter-Quartile Range); unit: mIU/L
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 52 | 54
mIU/L
  Pre-weight loss: number analyzed (Participants) | 56 | 51 | 54
  Pre-weight loss | 131.4 [77.6 to 173.5] | 116.7 [86.8 to 218.5] | 99.2 [73.7 to 153.4]
  Start of trial | 95.9 [55.5 to 131.3] | 79.9 [56.1 to 143.3] | 68.0 [57.0 to 106.6]
  End of test phase: number analyzed (Participants) | 53 | 48 | 45
  End of test phase | 96.2 [50.5 to 134.0] | 74.5 [51.3 to 135.4] | 74.8 [53.1 to 109.9]

30. Secondary Outcome: Thyroxine (T4)
Description: thyroid function test
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
nmol/L
  Pre-weight loss | 85 [78 to 95] | 86 [78 to 97] | 90 [79 to 102]
  Start of trial | 84 [75 to 96] | 85 [80 to 93] | 86 [78 to 96]
  End of test phase | 85 [78 to 94] | 86 [80 to 98] | 85 [77 to 98]

31. Secondary Outcome: Free T4
Description: free thyroxine, thyroid function test
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
pmol/L
  Pre-weight loss | 14.3 [13.1 to 15.9] | 15.0 [13.9 to 16.4] | 14.8 [13.5 to 16.1]
  Start of trial | 14.9 [13.6 to 15.9] | 15.2 [15.0 to 16.9] | 15.0 [14.1 to 15.8]
  End of test phase | 15.4 [14.0 to 16.6] | 15.7 [14.7 to 17.2] | 15.2 [14.0 to 16.1]

32. Secondary Outcome: Thyroid Stimulating Hormone
Description: Produced by the pituitary gland in the brain. Tells the thyroid gland to make thyroid hormones.
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: ulU/ml
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
ulU/ml
  Pre-weight loss | 2.0 [1.6 to 2.6] | 1.8 [1.4 to 2.5] | 2.1 [1.3 to 3.2]
  Start of trial | 2.1 [1.5 to 2.9] | 2.2 [1.5 to 2.7] | 2.5 [1.7 to 3.0]
  End of test phase | 2.0 [1.5 to 2.5] | 1.7 [1.4 to 2.7] | 2.1 [1.4 to 3.5]

33. Secondary Outcome: Reverse T3
Description: thyroid function test, inactive form of triiodothyronine (T3) Lifespan Bio kit was used for analysis. The range of this kit is 250 to 5000 pg/mL, which varies from other commercially available kits (about 10-fold greater values).
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers minus 1 participant in the High carbohydrate diet group for whom reverse T3 result is missing)
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 45
pg/mL
  Pre-weight loss | 1499 [1306 to 1610] | 1548 [1429 to 1676] | 1536 [1410 to 1756]
  Start of trial | 1545 [1356 to 1687] | 1554 [1383 to 1768] | 1548 [1378 to 1733]
  End of test phase | 1557 [1375 to 1702] | 1572 [1404 to 1795] | 1546 [1332 to 1686]

34. Secondary Outcome: Urinary Cortisol Excretion
Description: cortisol (stress hormone) excreted in the urine over a 24-hour period
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: μg/d
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
μg/d
  Pre-weight loss | 61 [48 to 78] | 59 [41 to 80] | 63 [45 to 91]
  Start of trial | 66 [48 to 83] | 64 [47 to 88] | 63 [50 to 77]
  End of test phase | 78 [56 to 100] | 64 [50 to 94] | 64 [45 to 84]

35. Secondary Outcome: Urinary Catecholamine - Adrenaline
Description: catecholamine excreted in the urine over 24 hours, also known as epinephrine
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: mcg/day
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
mcg/day
  Pre-weight loss | 3.1 [2.4 to 4.1] | 3.0 [2.2 to 4.2] | 2.9 [2.2 to 3.6]
  Start of trial | 3.5 [2.7 to 4.7] | 3.2 [2.3 to 4.3] | 3.0 [2.2 to 3.5]
  End of test phase | 3.6 [2.6 to 5.3] | 3.4 [2.3 to 4.7] | 3.1 [2.3 to 4.1]

36. Secondary Outcome: Urinary Catecholamine - Dopamine
Description: catecholamine excreted in the urine over 24 hours
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: mcg/day
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
mcg/day
  Pre-weight loss | 142.0 [105.7 to 187.5] | 143.2 [83.2 to 187.8] | 117.8 [92.7 to 163.6]
  Start of trial | 112.9 [75.1 to 157.6] | 112.4 [85.7 to 135.3] | 104.7 [76.0 to 125.9]
  End of test phase | 123.0 [86.4 to 159.1] | 112.9 [90.5 to 156.6] | 104.7 [83.9 to 141.7]

37. Secondary Outcome: Urinary Catecholamine - Noradrenaline
Description: catecholamine excreted in the urine over 24 hours, also known as norepinephrine
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: Descriptive data, reflecting participant flow End of test phase (N=148, completers)
Measure: Median (Inter-Quartile Range); unit: mcg/day
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 54 | 48 | 46
mcg/day
  Pre-weight loss | 25.8 [18.9 to 34.2] | 23.9 [18.9 to 31.6] | 25.3 [19.8 to 31.1]
  Start of trial | 25.2 [19.4 to 31.6] | 25.3 [20.1 to 31.7] | 24.7 [17.5 to 30.5]
  End of test phase | 27.4 [18.8 to 36.1] | 26.1 [20.6 to 36.9] | 26.0 [19.5 to 32.4]

38. Secondary Outcome: Insulin Sensitivity (Hepatic), Assessed by Frequently-sampled Oral Glucose Tolerance Test
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

39. Secondary Outcome: Insulin Sensitivity (Systemic), Assessed by Frequently-sampled Oral Glucose Tolerance Test
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

40. Secondary Outcome: Non-esterified Fatty Acids
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

41. Secondary Outcome: Serum Ketones/Ketoacids
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

42. Secondary Outcome: Lactate
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

43. Secondary Outcome: Metabolic Fuel Concentration in Serum (Glucose, Nonesterified Fatty Acids, Ketones/Ketoacids, Lactate)
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

44. Secondary Outcome: Insulin-like Growth Factor 1 (IGF-1)
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

45. Secondary Outcome: IGF Binding Proteins
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

46. Secondary Outcome: Testosterone
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

47. Secondary Outcome: Estradiol
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

48. Secondary Outcome: Luteinizing Hormone
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

49. Secondary Outcome: Follicle Stimulating Hormone
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

50. Secondary Outcome: Body Weight Change During ad Libitum Feeding
Time Frame: Ad libitum feeding period (weeks 21 and 22 following randomization)
Reporting Status: Not Posted, anticipated posting 2026-12

51. Secondary Outcome: Gut Microbiome Profile
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

52. Secondary Outcome: Serum Metabolomics Profile
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

53. Secondary Outcome: Change in Cognitive Function Related to Memory
Description: California Verbal Learning Test - Second Edition [CVLT-II] and Digit Span Test
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

54. Secondary Outcome: Change in Cognitive Function Related to Processing Speed and Executive Function
Description: Trail Making Test Parts A and B [TMT-A, TMT-B]
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

55. Secondary Outcome: Change in Self-reported Sleep Quality
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

56. Secondary Outcome: Change in Self-reported Depression Measure
Description: Beck Depression Inventory-II [BDI-II]
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

57. Secondary Outcome: Change in Self-reported Mood/Anxiety
Description: Mood and Anxiety Symptom Questionnaire [MASQ]
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

58. Secondary Outcome: Change in Self-reported Food Addiction Score
Description: Yale Food Addiction Scale [YFAS]
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

59. Secondary Outcome: Change in Self-reported Emotional Eating Score
Description: Emotional Eating Scale [EES]
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

60. Secondary Outcome: Change in Self-reported Binge Eating Score
Description: Binge Eating Scale [BES]
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

61. Other Pre Specified Outcome: Effect Modification by Insulin Secretion of Metabolic Responses to Diet
Description: Effect modifier: Insulin level 30 minutes into an standard OGTT (Insulin-30) Outcome: Total Energy Expenditure Tertiles: Pre-weight-loss Insulin-30 (Low, Moderate, High) Change: average (midpoint of test phase, end of test phase) - start of trial
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Population: The outcome is "Effect Modification by Insulin Secretion." Thus,participants were divided into tertiles of Insulin-30.
  Tertile I: Low=17, Moderate=16, High=22 Tertile II: Low=15, Moderate=22, High=17 Tertile III: Low=24, Moderate=14, High=15
Measure: Mean (95% Confidence Interval); unit: kcal/d
Arm/Group | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
Number analyzed (Participants) | 56 | 52 | 54
kcal/d
  Start of Trial, Low Insulin-30: number analyzed (Participants) | 17 | 16 | 22
  Start of Trial, Low Insulin-30 | 2795 [2591 to 2998] | 2673 [2456 to 2891] | 2647 [2463 to 2832]
  Change, Low Insulin-30: number analyzed (Participants) | 17 | 16 | 22
  Change, Low Insulin-30 | 147 [-1 to 295] | 103 [-44 to 250] | 15 [-119 to 148]
  Start of Trial, Moderate Insulin-30: number analyzed (Participants) | 15 | 22 | 17
  Start of Trial, Moderate Insulin-30 | 2816 [2597 to 3035] | 2563 [2377 to 2750] | 2782 [2571 to 2993]
  Change, Moderate Insulin-30: number analyzed (Participants) | 15 | 22 | 17
  Change, Moderate Insulin-30 | 114 [-37 to 266] | -5 [-136 to 127] | -50 [-200 to 101]
  Start of Trial, High Insulin-30: number analyzed (Participants) | 24 | 14 | 15
  Start of Trial, High Insulin-30 | 2643 [2461 to 2826] | 2281 [2053 to 2508] | 2544 [2331 to 2757]
  Change, High Insulin-30: number analyzed (Participants) | 24 | 14 | 15
  Change, High Insulin-30 | 271 [145 to 396] | 141 [-20 to 303] | -37 [-201 to 127]

62. Other Pre Specified Outcome: Effect Modification by Insulin Resistance of Metabolic Responses to Diet
Time Frame: Start of (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

63. Other Pre Specified Outcome: Effect Modification by Amylase Gene Copy Number
Time Frame: Start of trial (time of randomization, post-weight loss) through 20 weeks' weight loss maintenance
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the run-in diet (~12 weeks) and the test diet (20 weeks) periods of the study, a total of ~32 weeks.
Groups:
- Run-in Phase: Pre-randomization: During the run-in phase, energy intake was restricted to promote 12% (within 2%) weight loss over 9-10 weeks.
- Low Carbohydrate Diet: Feeding study: Composition (by proportion of calories): 20% carbohydrate, 60% fat, 20% protein.
- Moderate Carbohydrate Diet: Feeding study: Composition (by proportion of calories): 40% carbohydrate, 40% fat, 20% protein.
- High Carbohydrate Diet: Feeding study: Composition (by proportion of calories): 60% carbohydrate, 20% fat, 20% protein
Arm/Group | Run-in Phase | Low Carbohydrate Diet | Moderate Carbohydrate Diet | High Carbohydrate Diet
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/57 | 0/53 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/234 | 0/57 | 0/53 | 2/54
Other Adverse Events (participants affected / at risk) | 28/234 | 5/57 | 6/53 | 1/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase (N=234) | Low Carbohydrate Diet (N=57) | Moderate Carbohydrate Diet (N=53) | High Carbohydrate Diet (N=54)
Laparoscopic cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Removal of intrauterine device (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase (N=234) | Low Carbohydrate Diet (N=57) | Moderate Carbohydrate Diet (N=53) | High Carbohydrate Diet (N=54)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy, aversion or intolerance (Immune system disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood changes (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased blood cholesterol (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Possible gall bladder disease (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Possible hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Vomiting (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
High blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tested to rule out meningitis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Possible post-viral lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (new prescription medication) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study has three main limitations: potential measurement error, non-compliance, and generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT02068885/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT02068885/SAP_000.pdf